CLINICAL TRIAL: NCT04964869
Title: Efficacy of Prophylactic Epinephrine Solution Injection in Prevention of Delayed Post-sphincterotomy Bleeding in Patients with Transient Bleeding During ERCP
Brief Title: Efficacy of Prophylactic Epinephrine Solution Injection in Prevention of Delayed Post-sphincterotomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wen-Hsin Huang (Other)
Responsible Party: Sponsor-Investigator, Wen-Hsin Huang, Gastroenterology and Hepatology Deputy Director, China Medical University Hospital
Organization: China Medical University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CMUH110-REC2-055
Record Dates: First submitted 2021-07-08; First posted 2021-07-16 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Bleeding Hemorrhage
Keywords: sphincterotomy; epinephrine solution
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Epinephrine solution injection group (Experimental): In injected group, The saline epinephrine solution (1mg in 10ml N/S) is injected to 2 sites of cutted papilla (1 o'clock and 11 o'clock) by injected needle, at least 0.5ml per injected site, and must be protruded from submucosal layer.
  Interventions: Procedure: epinephrine solution injection
- non-injection group (No Intervention): In non injection group, the saline epinephrine solution is not given

INTERVENTIONS:
Procedure: epinephrine solution injection — epinephrine solution injection at least 1 ml to the post- sphincterotomy wound
  Arms: Epinephrine solution injection group

SUMMARY:
Bleeding is the most frequently reported serious complication of endoscopic sphincterotomy, and severe bleeding has occurred in about 1% to 2% of patients. Endoscopic injection of epinephrine is the most commonly used, effective, and least expensive method for the management of post- sphincterotomy bleeding. However, the efficacy of prophylactic saline-epinephrine solution injection to prevent delayed EST bleeding when transient bleeding During ERCP has not been established.

DETAILED DESCRIPTION:
Backgroud:

Bleeding is the most frequently reported serious complication of endoscopic sphincterotomy, and severe bleeding has occurred in about 1% to 2% of patients. Endoscopic injection of epinephrine is the most commonly used, effective, and least expensive method for the management of post- sphincterotomy bleeding. However, the efficacy of prophylactic saline-epinephrine solution injection to prevent delayed EST bleeding when transient bleeding During ERCP has not been established.

Study Rationale:

The hypotheses of the study is the prophylactic saline-epinephrine solution injection affects incidence of delayed post-EST bleeding.

Study Design:

A single blinded parallel group, multiple center, randomized controlled trial. The sample size is estimated 400 (200 in injection group and 200 in non-injection group), The primary outcome is the rate of delayed EST bleeding within 30 days of ERCP.

Study Objectives:

Primary objective: the rate of post-EST bleeding within 30 days of ERCP Secondary objectives: the rate of post-ERCP advese effect, the increasing procedure time because of hemostasis, the need for angiographic/endoscopic hemostasis times.

ELIGIBILITY:
Inclusion Criteria:

* Age 20 years or older.
* Ability to give informed consent.
* An naive major papilla.
* Transient bleeding after endoscopic sphincterotomy
* Bleeding less than 30 secs when end of procedure

Exclusion Criteria:

* Prior endoscopic sphincterotomy.
* Thrombocytopenia (platelets <50,000/mm3).
* Liver cirrhosis (Child A-C)
* CKD stage 4-5 and dialysis.
* Allergy to epinephrine
* Prolonged PT/APTT (INR>1.5)
* Had exposure any antithrombotic or antiplatelet agent in recent 7 days and/or will take those agents in one month after EST
* Ampulla Vater tumor
* Active GI bleeding
* Pregnancy
* Limited visibility when immediate bleeding after sphincterotomy
* Still bleeding after 30 secs when end of procedure
* Recurrent bleeding during ERCP

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2021-07-15 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
post EST bleeding rate | 30 days
  delay post-sphincterotomy bleeding rate

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Hsin Huang, MD, Principal Investigator — China Medical University Hospital
Locations (1):
- China Medical University Hospital, Taichung, North Dist., Taiwan